CLINICAL TRIAL: NCT03440164
Title: Superior Bioavailability of the Silybin-Phosphatidylcholine Complex in Oily-Medium Soft-Gel Capsules Versus Conventional Silymarin Tablets in Healthy Volunteers
Brief Title: Superior Silybin Bioavailability in Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: Medica Sur Clinic & Foundation (Other)
Responsible Party: Principal Investigator, Nahum Méndez-Sánchez, Gastroenterologist and Hepatologist, Medica Sur Clinic & Foundation
Other Study IDs: CONBIOETICA14CEI02820131108
Record Dates: First submitted 2018-02-14; First posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2016-10

CONDITIONS: Liver Diseases; Chronic Liver Disease
Keywords: liver fibrosis; Hepatoprotective; Sylimarin
MeSH Terms: conditions — Liver Diseases; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Sylimarin and Sylibin — We compared the plasma levels of Silibinin after a dosage of Silibinin-phosphatidylcholine complex, equivalent to 45 mg Silybin oily-medium soft-gel capsules after the conventional 70-mg Silymarin tablets, in 23 healthy volunteers

SUMMARY:
Twenty-four healthy volunteers of both genders, aged 18 to 44 years old and body mass indexes between 18 to 27 kg/m2,were selected to participate in a two-way, balanced, prospective, blind, single-dose crossover study with a one-week wash-out period. It was assessed that volunteers were free from significant cardiac, hepatic, renal, pulmonary, neurological, gastrointestinal and hematological diseases. The volunteers clinical evaluation were determined by clinical examination, ECG, and the following laboratory tests: blood glucose, urea, creatinine, AST, ALT, GGT, alkaline phosphatase, total bilirubin and fractions, uric acid, total cholesterol, triglycerides, albumin and total protein, and routine urinalysis. All subjects were negative for HIV, HBV, and HCV.

DETAILED DESCRIPTION:
In healthy volunteers single-dose crossover study with a one week, It was assessed that volunteers were free from significant cardiac, hepatic, renal, pulmonary, neurological, gastrointestinal and hematological diseases. The volunteers clinical evaluation were determined by clinical examination

ELIGIBILITY:
Inclusion Criteria:

* volunteers were free from significant cardiac, hepatic, renal, pulmonary, neurological, gastrointestinal and hematological diseases.

The volunteers clinical evaluation were determined by clinical examination, ECG, and the following laboratory tests: blood glucose, urea, creatinine, AST, ALT, GGT, alkaline phosphatase, total bilirubin and fractions, uric acid, total cholesterol, triglycerides, albumin and total protein, and routine urinalysis

Exclusion Criteria:

* Subject with HIV, HBV, HCV
* Subject with comorbidities
* Subject less 18 years old Subject higher 50 years old

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: All healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2016-11-11 (Actual); Primary Completion 2016-12-08 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
Time of the Bioavailability of the Silibinin vs Sylimarin | One week
  Analysis of the Bioavailability

IPD SHARING:
Plan to Share IPD: Yes
Our results will be published in a scientific journal
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: From 2017 to date
Access Criteria: Publication in Open Acess

REFERENCES:
- [Derived] Mendez-Sanchez N, Dibildox-Martinez M, Sosa-Noguera J, Sanchez-Medal R, Flores-Murrieta FJ. Superior silybin bioavailability of silybin-phosphatidylcholine complex in oily-medium soft-gel capsules versus conventional silymarin tablets in healthy volunteers. BMC Pharmacol Toxicol. 2019 Jan 11;20(1):5. doi: 10.1186/s40360-018-0280-8. PMID 30635055